CLINICAL TRIAL: NCT00427882
Title: An Open, Non-Comparative, Multicenter Study on the Sexual Function Improvement Following Treatment With Alfuzosin in Patients With Benign Prostate Hyperplasia
Brief Title: Male Sexual Health Questionnaire (MSHQ) - Sexual Function Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALFUS_L_01778
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

INTERVENTIONS:
Drug: ALFUZOSIN

SUMMARY:
Primary:

To assess improvement in ejaculation from baseline to the end of treatment (Week 12 or premature withdrawal) with Alfuzosin 10mg OD, using MSHQ score.

Secondary:

* To evaluate sexual function improvement
* To evaluate LUTS (Lower Uninary Tract Symptoms) improvement
* To evaluate the association between LUTS severity and sexual function.
* To assess the safety and the tolerability of Alfuzosin 10mg OD.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from moderate to severe lower urinary tract symptoms (LUTS), suggestive of symptomatic Benign Prostatic Hyperplasia (BPH) diagnosed by the Investigator
* Patients with an I-PSS total score ≥ 8
* Patients sexually active as defined by at least one of the following activities in the last 4 weeks: intercourse, caressing, foreplay, masturbation

Exclusion Criteria:

* Patients with a known history of hepatic or severe renal insufficiency, unstable angina pectoris
* Patients who had a previous prostate surgery
* Patients who had a prostate biopsy or minimally invasive procedure within 6 months prior to inclusion
* Patients with a prostate surgery or minimally invasive procedure during the whole study period
* Patients with an active urinary tract infection or prostatitis
* Patients with a neuropathic bladder defined as a spinal injury consequence or related to a neurological disorder or a known residual volume ≥ 350 ml
* Patients with a diagnosed prostate cancer
* Patients having received 5a-reductase inhibitors or LUTS related-phytotherapy within 6 months prior to inclusion, or a1-blockers within 30 days prior to inclusion
* Patients receiving any treatment for erectile dysfunction (i.e. phosphodiesterase-5 inhibitors) at inclusion
* Patients with a history of postural hypotension or syncope
* Patients with a known hypersensitivity to alfuzosin

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2006-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to the end of treatment in the MSHQ ejaculation total score

SECONDARY OUTCOMES:
Mean change from baseline to 4 weeks in MSHQ ejaculation total score
Mean change from baseline to 4 weeks and the end of treatment in MSHQ erection total score and in the satisfaction total score
Mean change from baseline to 4 weeks and the end of treatment in MSHQ ejaculation questions, in the erection and satisfaction sub-scores
Mean change from baseline to 4 weeks and the end of treatment in the I-PSS (International Prostate Symptom Score) total score and in the Quality of Life
Mean change from baseline to 4 weeks and the end of treatment in I-PSS sub-scores for voiding, filling and nocturia symptoms
Mean change from baseline to 4 weeks and the end of treatment in the peak urinary flow rate (Qmax)
Correlation between MSHQ and IPSS
Evaluation of adverse events, vital signs (blood pressure and heart rate in sitting position), PSA (Prostate Specific Antigen) and creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Hyou-Young Rhim, Dr., Study Director — Handok Inc.
Locations (1):
- Handok, Seoul, South Korea